CLINICAL TRIAL: NCT04178824
Title: Multi-level Supermarket Discounts of Fruits and Vegetables' Impact on Intake and Health
Brief Title: Multi-level Supermarket Discount Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Allan Geliebter, Professor, Department of Psychiatry, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 16-1050; R01DK105440 (NIH)
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Obesity
Keywords: Nutrition
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 15% discount intervention (Experimental): 15% discount on fruits, vegetables and non-caloric beverages at the designated supermarkets
  Interventions: Behavioral: Discount Intervention
- Experimental 30% discount intervention (Experimental): 30% discount on fruits, vegetables and non-caloric beverages at the designated supermarkets
  Interventions: Behavioral: Discount Intervention
- No intervention control group (No Intervention): 0% discount on fruits, vegetables and non-caloric beverages at the designated supermarkets

INTERVENTIONS:
Behavioral: Discount Intervention — 15% or 30% discount on fruits and vegetables
  Arms: Experimental 15% discount intervention; Experimental 30% discount intervention

SUMMARY:
The study team's objective is to test the effect of supermarket discount levels on fruit and vegetable (F&V) and non-caloric beverage purchasing and consumption, as well as health outcomes. The study team will implement this economic intervention in a local supermarket chain to assess the effects of a 32-week intervention of fruit and vegetable (F&V) and non-caloric beverage discounts of 30%, 15%, and 0% (control group) on purchasing, dietary intake, and health outcomes, including body weight and composition, blood pressure, and biochemical markers of cardiovascular disease risk. The 32-week intervention will be preceded by an 8-week baseline and will have a follow-up period of 16 weeks. There will be no discounts in effect during the baseline and follow-up periods.

DETAILED DESCRIPTION:
The objective is to test the effect of supermarket discount levels on fruit and vegetable (F&V) and non-caloric beverage purchasing and consumption, as well as health outcomes. The study team will implement this economic intervention in a local supermarket chain to assess the effects of a 32-week intervention of fruit and vegetable (F&V) and non-caloric beverage discounts of 30%, 15%, and 0% (control group) on purchasing, dietary intake, and health outcomes, including body weight and composition, blood pressure, and biochemical markers of cardiovascular disease risk. The prediction is that the impact will increase with the level of discount. The 32-week intervention will be preceded by an 8-week baseline and will have a follow-up period of 16 weeks. There will be no discounts in effect during the baseline and follow-up periods. The prediction is that some of the interventional effects will carry over to the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 24.5 - 50
* Weight Stable (±5% body weight in last 3 mo)
* Accessible by telephone
* Living in NYC and not planning move
* Primary household food shopper
* ≥50% of food shopping at Foodtown/Brooklyn Harvest and agrees to 100% shopping at store during study
* Consumption of >50% of food shopping
* Eat out or take out ≤5 times weekly

Exclusion Criteria:

* Pregnant or contemplating pregnancy
* Enrolled in related studies
* Active weight loss program
* Presence of serious medical (e.g. cancer, diabetes) or psychiatric disease (e.g. bipolar)
* Changes in medications or smoking in past 3 mo
* Excessive alcohol use (≥4 drinks/day) or illicit drug use
* Planning a vacation ≥ 4 consecutive weeks or 6 total weeks during study
* Receiving SNAP benefits

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Geliebter, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai St. Luke's, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available upon request after study completion and publication.
Supporting Information: Study Protocol, CSR
Time Frame: Data should become available 12/23
Access Criteria: Can be requested of the PI by other investigators.

REFERENCES:
- [Result] Poskute AS, Nzesi A, Geliebter A. Changes in food intake during the COVID-19 pandemic in New York City. Appetite. 2021 Aug 1;163:105191. doi: 10.1016/j.appet.2021.105191. Epub 2021 Mar 3. PMID 33667497
- [Result] Nzesi A, Roychowdhury L, De Jesus ML, Brown A, Geliebter A. Body weight, dietary intake, and health risk factors pre-COVID and during the COVID-19 pandemic. Appetite. 2022 Nov 1;178:106182. doi: 10.1016/j.appet.2022.106182. Epub 2022 Aug 6. PMID 35940334
- [Result] Nzesi A, Owusu B, Barry J, Sandhu M, Geliebter A. Impact of a randomized controlled trial of discounts on fruits, vegetables, and noncaloric beverages in NYC supermarkets on food intake and health risk factors. PLoS One. 2023 Nov 22;18(11):e0291770. doi: 10.1371/journal.pone.0291770. eCollection 2023. PMID 37992046
- [Result] Poskute AS, Ang IYH, Rahman N, Geliebter A. Effects of discounting fruits, vegetables, and noncaloric beverages in New York City supermarkets on purchasing, intake, and weight. Obesity (Silver Spring). 2024 Jul;32(7):1290-1301. doi: 10.1002/oby.24058. PMID 38932711

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Started | 57 | 57 | 53
Completed | 38 | 33 | 36
Not Completed | 19 | 24 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group | Total
Number analyzed (Participants) | 38 | 33 | 36 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (12.9) | 41.8 (14.3) | 39.6 (11.7) | 40.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 24 | 67
  Male | 14 | 14 | 12 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 6 | 20
  Not Hispanic or Latino | 28 | 25 | 24 | 77
  Unknown or Not Reported | 2 | 2 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 2 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 11 | 7 | 17 | 35
  White | 21 | 15 | 8 | 44
  More than one race | 2 | 2 | 1 | 5
  Unknown or Not Reported | 3 | 6 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Fruit Intake as Assessed by 24-h Dietary Recalls
Description: Individual consumption behaviors: Fruit intake as assessed by 24-h dietary recalls
Time Frame: Week 8, 24, 40, 56
Measure: Mean (95% Confidence Interval); unit: grams
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 38 | 33 | 36
grams
  Week 8 | 99.6 [57.1 to 142] | 112 [66.6 to 157] | 93.4 [49.6 to 137]
  Week 24 | 127 [84.5 to 169] | 120 [75.3 to 166] | 112 [67.8 to 155]
  Week 40 | 105 [60 to 149] | 137 [90.5 to 183] | 86.8 [40.4 to 133]
  Week 56 | 198 [149 to 248] | 124 [76.5 to 171] | 54.9 [3.35 to 106]

2. Primary Outcome: Vegetable Intake as Assessed by 24-h Dietary Recalls
Description: Individual consumption behaviors: Vegetable intake as assessed by 24-h dietary recalls
Time Frame: Week 8, 24, 40, 56
Measure: Mean (95% Confidence Interval); unit: grams
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 38 | 33 | 36
grams
  Week 8 | 185 [137 to 232] | 126 [75.3 to 176] | 158 [110 to 207]
  Week 24 | 190 [143 to 237] | 192 [142 to 242] | 136 [87.6 to 185]
  Week 40 | 163 [114 to 213] | 175 [123 to 227] | 152 [100 to 204]
  Week 56 | 137 [81.4 to 193] | 157 [104 to 210] | 176 [119 to 234]

3. Primary Outcome: Bottled Water Intake as Assessed by 24-h Dietary Recalls
Description: Individual consumption behaviors: bottled water intake as assessed by 24-h dietary recalls
Time Frame: Week 8, 24, 40, 56
Measure: Mean (95% Confidence Interval); unit: grams
Groups:
- Experimental 30% Discount Intervention: 30% discount on fruits, vegetables and non-caloric beverages at the designated supermarket
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 38 | 33 | 36
grams
  Week 8 | 93 [-47.9 to 234] | 178 [28.5 to 328] | 132 [-13.2 to 277]
  Week 24 | 137 [-2.55 to 276] | 156 [6.59 to 306] | 190 [44.8 to 334]
  Week 40 | 217 [69.3 to 365] | 202 [48.6 to 355] | 272 [118 to 427]
  Week 56 | 179 [13.3 to 345] | 86.8 [-70.9 to 244] | 264 [91.5 to 437]

4. Primary Outcome: Seltzer Water Intake as Assessed by 24-h Dietary Recalls
Description: Individual consumption behaviors: seltzer water intake as assessed by 24-h dietary recalls
Time Frame: Week 8, 24, 40, 56
Measure: Mean (95% Confidence Interval); unit: grams
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 38 | 33 | 36
grams
  Week 8 | 50.4 [-26.4 to 127] | 47.9 [-33.9 to 130] | 134 [54.7 to 213]
  Week 24 | 64.4 [-11.8 to 141] | 65.2 [-16.6 to 147] | 157 [78.2 to 236]
  Week 40 | 77.6 [-2.49 to 158] | 21.3 [-62.2 to 105] | 159 [75.3 to 242]
  Week 56 | 61.6 [-26.9 to 150] | 84.8 [-0.702 to 170] | 182 [90 to 274]

5. Primary Outcome: Diet Soda Intake as Assessed by 24-h Dietary Recalls
Description: Individual consumption behaviors: diet soda intake as assessed by 24-h dietary recalls
Time Frame: Week 8, 24, 40, 56
Measure: Mean (95% Confidence Interval); unit: grams
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 38 | 33 | 36
grams
  Week 8 | 1.89 [-35.5 to 39.3] | 33.6 [-6.34 to 73.6] | 37.5 [-1 to 75.9]
  Week 24 | 12.5 [-24.8 to 49.7] | 78.9 [38.9 to 119] | 15.1 [-23.3 to 53.6]
  Week 40 | 4.19 [-34.1 to 42.4] | 57.5 [17.1 to 98] | 18.9 [-20.7 to 58.5]
  Week 56 | 13.2 [-27.1 to 53.6] | 69.1 [28.2 to 110] | 16.3 [-25.5 to 58]

6. Primary Outcome: Total Non-caloric Beverage Intake as Assessed by 24-h Dietary Recalls
Description: Individual consumption behaviors: Total non-caloric beverage intake as assessed by 24-h dietary recalls
Time Frame: Week 8, 24, 40, 56
Measure: Mean (95% Confidence Interval); unit: grams
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 38 | 33 | 36
grams
  Week 8 | 146 [-14.6 to 306] | 260 [89.5 to 430] | 304 [139 to 468]
  Week 24 | 213 [54.1 to 371] | 285 [115 to 455] | 362 [198 to 527]
  Week 40 | 299 [131 to 467] | 281 [107 to 456] | 450 [274 to 626]
  Week 56 | 253 [64.3 to 441] | 243 [64.2 to 422] | 465 [269 to 661]

7. Secondary Outcome: Body Weight
Description: Body weight (kg)
Time Frame: Week 0, 8, 24, 40, 56
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 38 | 33 | 36
kilograms
  Week 0 | 84 [78.4 to 89.7] | 83.5 [77.5 to 89.5] | 83.3 [77.5 to 89.1]
  Week 8 | 84.3 [78.6 to 89.9] | 82.8 [76.8 to 88.8] | 84.6 [78.8 to 90.4]
  Week 24 | 84.4 [78.8 to 90] | 83 [77 to 89] | 85.2 [79.4 to 91]
  Week 40 | 84.2 [78.5 to 89.8] | 83.9 [77.8 to 89.9] | 84.6 [78.8 to 90.5]
  Week 56 | 86 [80.3 to 91.6] | 83.4 [77.4 to 89.5] | 84.3 [78.5 to 90.1]

8. Secondary Outcome: Body Mass Index (BMI)
Description: BMI (kg/m^2)
Time Frame: Week 0, 8, 24, 40, 56
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 38 | 33 | 36
kg/m^2
  Week 0 | 29.7 [27.8 to 31.5] | 29.7 [27.7 to 31.6] | 29.3 [27.4 to 31.2]
  Week 8 | 29.7 [27.8 to 31.5] | 29.5 [27.5 to 31.4] | 29.6 [27.8 to 31.5]
  Week 24 | 29.8 [28 to 31.6] | 29.1 [27.1 to 31] | 29.9 [28.1 to 31.8]
  Week 40 | 29.7 [27.9 to 31.6] | 29.8 [27.8 to 31.8] | 29.6 [27.7 to 31.5]
  Week 56 | 29.8 [27.9 to 31.6] | 29.6 [27.6 to 31.6] | 29.6 [27.7 to 31.6]

9. Secondary Outcome: Percent Body Fat
Description: % body fat
Time Frame: Week 0, 8, 24, 40, 56
Measure: Mean (95% Confidence Interval); unit: percent of body fat
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 38 | 33 | 36
percent of body fat
  Week 0 | 34 [30.7 to 37.4] | 33.2 [29.6 to 36.8] | 33.4 [30 to 36.9]
  Week 8 | 33.5 [30.1 to 36.8] | 32.6 [29 to 36.2] | 33.3 [29.9 to 36.7]
  Week 24 | 34 [30.7 to 37.4] | 33 [29.4 to 36.6] | 34.2 [30.8 to 37.7]
  Week 40 | 34.1 [30.7 to 37.5] | 33.8 [30.2 to 37.4] | 34.4 [30.9 to 37.9]
  Week 56 | 34.2 [30.8 to 37.6] | 33.5 [29.9 to 37.1] | 34.2 [30.7 to 37.7]

10. Secondary Outcome: Waist Circumference
Description: Waist circumference (cm)
Time Frame: Week 0, 8, 24, 40, 56
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 38 | 33 | 36
centimeters
  Week 0 | 37.9 [36.1 to 39.8] | 37.5 [35.5 to 39.5] | 38.3 [36.4 to 40.2]
  Week 8 | 38.3 [36.5 to 40.2] | 37.7 [35.7 to 39.7] | 38.6 [36.7 to 40.5]
  Week 24 | 38 [36.2 to 39.9] | 37.6 [35.6 to 39.5] | 37.6 [35.7 to 39.5]
  Week 40 | 37.7 [35.8 to 39.6] | 37.5 [35.5 to 39.4] | 38.3 [36.4 to 40.3]
  Week 56 | 38 [36.1 to 39.9] | 37.8 [35.8 to 39.7] | 37.6 [35.6 to 39.5]

11. Secondary Outcome: Fasting Glucose
Description: Fasting glucose level
Time Frame: Week 0, 8, 24, 40, 56
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 38 | 33 | 36
mg/dL
  Week 0 | 87.6 [83.8 to 91.5] | 87.4 [83.1 to 91.7] | 85 [80.9 to 89.2]
  Week 8 | 91.5 [87.6 to 95.4] | 91.5 [87.1 to 95.8] | 86.3 [82.3 to 90.3]
  Week 24 | 90.1 [86 to 94.1] | 93.1 [88.8 to 97.4] | 89.3 [85 to 93.7]
  Week 40 | 90.3 [85.3 to 95.3] | 89.7 [84.6 to 94.7] | 89.5 [84.7 to 94.4]
  Week 56 | 97.1 [92 to 102] | 96.9 [92 to 102] | 91.1 [85.8 to 96.3]

12. Secondary Outcome: Cholesterol Level
Description: Cholesterol level
Time Frame: Week 0, 8, 24, 40, 56
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 38 | 33 | 36
mg/dL
  Week 0 | 182 [171 to 192] | 184 [173 to 196] | 192 [181 to 203]
  Week 8 | 173 [162 to 183] | 183 [172 to 194] | 194 [183 to 204]
  Week 24 | 183 [172 to 193] | 183 [172 to 194] | 196 [185 to 207]
  Week 40 | 180 [169 to 192] | 180 [169 to 192] | 190 [179 to 202]
  Week 56 | 182 [171 to 193] | 188 [177 to 200] | 198 [187 to 210]

13. Secondary Outcome: Blood Pressure
Description: Blood pressure systolic and diastolic.
Time Frame: Week 0, 8, 24, 40, 56
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 38 | 33 | 36
mmHg
  Week 0 systolic | 121 [116 to 125] | 117 [112 to 122] | 122 [117 to 127]
  Week 0 diastolic | 76.1 [73.4 to 78.9] | 73 [70.1 to 75.9] | 77.7 [74.9 to 80.5]
  Week 8 systolic | 120 [115 to 124] | 115 [110 to 120] | 121 [117 to 126]
  Week 8 diastolic | 75.6 [72.9 to 78.3] | 72.4 [69.4 to 75.4] | 78.3 [75.5 to 81.1]
  Week 24 systolic | 119 [114 to 123] | 116 [111 to 121] | 121 [116 to 126]
  Week 24 diastolic | 75 [72.3 to 77.7] | 71.7 [68.8 to 74.7] | 77.8 [75 to 80.6]
  Week 40 systolic | 116 [111 to 121] | 118 [113 to 123] | 122 [117 to 128]
  Week 40 diastolic | 75.1 [71.9 to 78.2] | 75.1 [72 to 78.2] | 75.2 [71.9 to 78.4]
  Week 56 systolic | 115 [110 to 121] | 117 [112 to 123] | 120 [114 to 126]
  Week 56 diastolic | 76 [72.8 to 79.1] | 74.1 [70.9 to 77.2] | 78.4 [75 to 81.7]

14. Secondary Outcome: Gross Weekly Purchasing of Fruits and Vegetables
Description: Gross weekly purchasing of fruits and vegetables from the discounted items list in dollars
Time Frame: Week 8-56
Population: Data was not collected as it was not received from vendor due to privacy concerns.
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 56 weeks
Arm/Group | Experimental 15% Discount Intervention | Experimental 30% Discount Intervention | No Intervention Control Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/33 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/33 | 0/36
Other Adverse Events (participants affected / at risk) | 0/38 | 0/33 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT04178824/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT04178824/SAP_001.pdf
  • Informed Consent Form (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT04178824/ICF_002.pdf